CLINICAL TRIAL: NCT05922943
Title: Harmony & Health: A Culturally Adapted Mindbody Intervention to Reduce Sitting Time and Improve Psychosocial Wellbeing in Black Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society (ACS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0321; NCI-2023-04992 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Psychosocial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Harmony & Health program (Experimental): Participants will take part in the Harmony & Health program or participants will attend in-person group health education sessions 2 times a week for 8 weeks.
  Interventions: Behavioral: Harmony & Health program

INTERVENTIONS:
Behavioral: Harmony & Health program — Harmony & Health program may help improve psychosocial wellbeing in participants and if improvements in physical activity and wellbeing can last after the program ends. Yoga combines gentle movements, breathing exercises, relaxation techniques, and meditation all tailored to the participant's needs.

SUMMARY:
This community-based study will assess the efficacy of a culturally adapted, yoga-based intervention to reduce sitting time, increase physical activity, and improve psychosocial wellbeing among insufficiently active Black adults in the Houston area.

DETAILED DESCRIPTION:
Primary Objectives:

--The primary aim of the proposed study is to determine the efficacy of HH in reducing sitting time and increasing physical activity in insufficiently active Black adults. Hypothesis: HH participants will spend less time sitting and more time moving at post-intervention (week 9) compared to participants in the attention control group.

Secondary Objectives:

The secondary aims of this proposed study are to:

* Examine the effects of HH on psychosocial wellbeing and the association of psychosocial wellbeing with behavioral outcomes. Hypothesis: HH participants will report improved psychosocial wellbeing, including reduced stress, depressive symptoms, and negative affect and improved quality of life, which will in turn mediate intervention outcomes at post-intervention (week 9) and follow up (week 24).
* Evaluate the long-term benefits of the HH intervention. Hypothesis: HH participants will spend less time sitting and more time moving at follow up (week 24) compared to participants in the attention control group.

An exploratory aim of the proposed study is to identify implementation facilitators and barriers using a mixed-methods approach. Implementation of HH will be evaluated using the Consolidated Framework for Implementation Research (CFIR) and the RE-AIM Framework. In-depth interviews with key informants combined with administrative and questionnaire data will be used to identify critical facilitators and barriers for implementing HH and to evaluate reach, implementation, adoption, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old
2. Self-identify as Black or African American
3. Self-reports MVPA <150 minutes/week
4. Self-reports sedentary time ≥6 hours/ day
5. Body mass index [BMI] ≥25.0 kg/m2 based on self-reported height and weight (and verified at baseline)
6. Able to pass the modified Physical Activity Readiness Questionnaire (PAR-Q) or provide physician's clearance to participate
7. Willing to be randomized to intervention or control
8. Comfortable participating in group-based physical activity
9. Able to read, speak, and write in English
10. Able to provide written informed consent without assistance

Exclusion Criteria:

1. < 18 years old
2. Self-reports MVPA .150 minutes/week
3. Self-reports sedentary time <6 hours/day
4. Not classified as overweight or obese (BMI <25.0 kg/m2)
5. Absolute contraindications to unassisted physical activity (e.g. acute MI, orthopedic and musculoskeletal limitations)
6. Practicing yoga or enrolled in another program targeting physical activity, sedentary behavior, or weight loss in the last 6 months
7. Previously participated in Harmony & Health
8. Pregnant or planning to become pregnant in the next 6 months
9. Planning to move from the Houston area within the next 6 months

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaires | through study completion; an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Scherezade Mama, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org